CLINICAL TRIAL: NCT03687762
Title: Mechanisms of Psychosocial Treatments for Chronic Pain
Brief Title: Back on Track to Healthy Living Study
Acronym: BOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Rush University (Other); Medical University of South Carolina (Other); The University of Queensland (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mark Jensen, Professor, School of Medicine: Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003841; R01AT008559 (NIH)
Record Dates: First submitted 2018-08-13; First posted 2018-09-27 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
Keywords: chronic pain; mechanisms; cognitive therapy; mindfulness meditation; behavioral activation
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy; Mindfulness

STUDY DESIGN:
Intervention Model Description: A randomized, 3-group parallel design, 240-subject clinical trial to test the mechanisms of cognitive therapy, mindfulness meditation, and behavioral activation on individuals with chronic pain who endorse low back pain as a primary or secondary pain problem.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Therapy (CT) Condition (Active Comparator): Participants randomized to this arm will be taught to recognize the relationships between thoughts, feelings, behaviors, and pain. This technique will help participants: (1) identify negative or unrealistic automatic thoughts; (2) evaluate automatic thoughts for accuracy, identify sources of distorted thoughts, recognize the connection between automatic thoughts and emotional/physical shifts; (3) challenge negative, distorted automatic thoughts via "weighing the evidence"; (4) develop new realistic alternative cognitive appraisals; and (5) practice applying new rational appraisals and beliefs.
  Interventions: Behavioral: Cognitive Therapy (CT)
- Mindfulness Meditation (MM) Condition (Active Comparator): Participants randomized to this arm will receive training in mindfulness meditation, specifically Vipassana, which is the form of meditation typically implemented in mindfulness research. With this technique, the emphasis is placed upon developing focused attention on an object of awareness, e.g., the breath. This focus is then expanded to include a more open, non-judgmental monitoring of any sensory, emotional, or cognitive events.
  Interventions: Behavioral: Mindfulness Meditation (MM)
- Behavioral Activation (BA) Condition (Active Comparator): Participants randomized to this arm will be educated about the role of inactivity and behavioral avoidance in chronic pain and functioning. They will learn how to be aware of the activities they avoid because of pain, and how to set effective goals so that, step by step, they can start being more active and resume some activities they enjoyed in the past but are currently avoiding. Explanation and practice of a set of specific skills - including appropriate pacing skills - to facilitate an increase in appropriate activity level will be provided.
  Interventions: Behavioral: Behavioral Activation (BA)

INTERVENTIONS:
Behavioral: Cognitive Therapy (CT) — The cognitive-restructuring technique will be used to help participants recognize the relationships between thoughts, feelings, behaviors, and pain. This technique will help participants: (1) identify negative or unrealistic automatic thoughts; (2) evaluate automatic thoughts for accuracy, identify sources of distorted thoughts, recognize the connection between automatic thoughts and emotional/physical shifts; (3) challenge negative, distorted automatic thoughts via "weighing the evidence"; (4) develop new realistic alternative cognitive appraisals; and (5) practice applying new rational appraisals and beliefs.
  Arms: Cognitive Therapy (CT) Condition
Behavioral: Mindfulness Meditation (MM) — Participants will receive training in mindfulness meditation, specifically Vipassana, which is the form of meditation typically implemented in mindfulness research. With this technique, the emphasis is placed upon developing focused attention on an object of awareness, e.g., the breath. This focus is then expanded to include a more open, non-judgmental monitoring of any sensory, emotional, or cognitive events. A standard script will be implemented by the clinician, and participants will be seated in a comfortable yet alert position.
  Arms: Mindfulness Meditation (MM) Condition
Behavioral: Behavioral Activation (BA) — Participants will be educated about the role of inactivity and behavioral avoidance in chronic pain and functioning. They will learn how to be aware of the activities they avoid because of pain, and how to set effective goals so that, step by step, they can start being more active and resume some activities they enjoyed in the past but are currently avoiding. Explanation and practice of a set of specific skills - including appropriate pacing skills - to facilitate an increase in appropriate activity level will be provided.
  Arms: Behavioral Activation (BA) Condition

SUMMARY:
Chronic pain is a significant problem affecting millions of Americans. Research has shown that psychological treatments can help people with chronic pain manage their pain and improve their quality of life. Three common psychological treatments for chronic pain are Cognitive Therapy (CT), Mindfulness Meditation (MM), and Behavioral Activation (BA). While research has shown these treatments are helpful for people with chronic pain, there is little research explaining why these treatments are helpful. The purpose of this study is to understand the specific ways these treatments work. Increasing our understanding of how these treatments work will help researchers and clinicians improve treatments for people with chronic pain in the future. As a secondary aim, this study will also examine the post-treatment mechanisms that explain relapse, maintenance, and continued gains associated with these treatments. Treatment moderators will also be explored.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to evaluate the mechanisms of cognitive therapy (CT), mindfulness meditation (MM), and behavioral activation (BA) as treatments for individuals with chronic pain who endorse low back pain as a primary or secondary pain problem. Participants (240 individuals) will be randomly assigned to eight (8), 1.5 hour telehealth group sessions of (1) CT, (2) MM, or (3) BA. Mechanisms and outcomes will be assessed twice daily during 2-week baseline, 4-week treatment period, and 4-week post-treatment epoch via cue-elicited ecological momentary assessment (EMA); activity level will be monitored during these time epochs via daily monitoring with ActiGraph technology. Follow-up macro-level assessments will be conducted at 3- and 6-months post-treatment. The study will address two aims.

Primary Objective: The objective of the proposed research is to examine the mechanisms of cognitive therapy (CT), mindfulness meditation training (MM), and behavioral activation (BA) [Aim 1; Primary]. After ensuring that there is at least a small effect of time on early treatment changes in the three mechanism variables, researchers will determine the extent to which late-treatment improvement in primary outcome (pain interference) associated with CT, MM, and BA is predicted by early-treatment changes in cognitive content (i.e., pain catastrophizing), cognitive process (i.e., non-judgment), and/or activity level (i.e., ActiGraph "activity counts").

Hypothesis 1a: Early treatment changes in pain catastrophizing, non-judgment, and activity counts are significantly associated with late treatment improvements in pain interference.

Hypothesis 1b: The Shared Mechanisms Model hypothesizes that if changes in cognitive content, cognitive process, and activity levels are shared mechanisms across the three treatments, then treatment condition will have small and non-significant effects on early changes in the mechanism variables (i.e., the effects of the three treatments on the three mechanism variables will be similar; Shared Mechanisms Model).

Hypothesis 1c: The Specific Mechanisms Model hypothesizes that if changes in content, process, and activity level are mechanisms specific to CT, MM, and BA, respectively, then treatment condition will have a significant effect on early changes in the mechanism variables (i.e., the effects of the three treatments on the three mechanism variables will be different, with CT having the largest effects on early treatment decreases in catastrophizing, MM having the largest effects on early treatment increases in non-judgment, and BA having the largest effects on early treatment increases in activity level). Further, later improvement in the primary outcome will be predicted by different mechanism variables as a function of treatment condition; that is, late treatment changes in pain interference will be substantially and uniquely predicted by early treatment changes in: (1) cognitive content (i.e., pain catastrophizing) in CT but not in MM or BA; (2) cognitive process (i.e., non-judgment) in MM but not in CT or BA; and (3) activity level in BA but not in CT or MM, in addition to each mechanism variable significantly predicting the primary outcome (Specific Mechanisms Model).

Researchers also predict that change in the mechanism variables will precede and predict change in outcome, but not vice versa.

Secondary Objective: As a secondary aim, this study will also evaluate the post-treatment mechanisms that explain relapse, maintenance, and continued gains associated with these treatments [Aim 2; Secondary]. The Shared (Hypothesis 2a) and Specific (Hypothesis 2b) Mechanism models will also be applied to data collected via EMA and ActiGraph daily during the 4-weeks post-treatment to better understand the post-treatment mechanisms that underlie maintenance of gains and relapse.

Exploratory Objective: Test the Limit, Activate, and Enhance (LAE) moderation model. Specifically, to test if (1) higher baseline levels of catastrophizing are associated with a positive response to the CT intervention, (2) lower baseline levels of activity are associated with a positive response to BA, and (3) higher baseline levels of non-judgment are associated with a positive response to MM.

Primary and Secondary Endpoint: The primary endpoint researchers propose for the primary study aim (Aim 1) is the post-treatment pain interference score, operationalized as an average of pain interference ratings made on the twice-daily diaries during the first four days after treatment (i.e., Days 43-46). The endpoint for the secondary study aim (Aim 2) is the post-treatment score at 28 days follow-up, as operationalized as the average of days 67-70 of pain interference ratings on the diaries.

Design and Outcomes

A randomized, 3-group parallel design, 240-subject clinical trial to test the mechanisms of cognitive therapy, mindfulness meditation, and activation skills on individuals with chronic pain who endorse low back pain as a primary or secondary pain problem.

Interventions and Duration

Participants will be randomly assigned to eight (8) telehealth group sessions of (1) cognitive therapy (CT), (2) mindfulness meditation (MM), or (3) behavioral activation (BA). Treatment groups will meet, on average, twice per week over the Zoom videoconferencing platform. Each session will last for a duration of about 90 minutes. Proposed mechanisms and outcomes will be assessed twice daily during 2-week baseline, 4-week treatment period, and 4-week post-treatment epoch via cue-elicited ecological momentary assessment (EMA); activity level will be monitored during these time epochs via daily monitoring with ActiGraph technology. Macro-level assessments will be conducted at pre- and post-treatment and at 3- and 6-months post-treatment.

The total time involved in the study (excluding between session skills practice) is approximately 35-40 hours over an 8 to 9-month period.

Sample Size and Population

Researchers plan to enroll 300 participants with moderate to severe chronic pain including low back pain as a primary or secondary pain problem to achieve a sample size of 240 completers, with 80 completers in each of the treatment groups.

Enrolled participants who complete the required baseline components (baseline data and demographic questions, pre-treatment extended assessment period, technology training, re-assessment of pain interference for general activities with a score of ≥3 for the past 3 months, re-assessment of pain consistency with a response of ≥50% of the time in the past 6 months, and a minimum number of EMA surveys during one week of Baseline Monitoring (Days 1-7) will be randomized to one of the three conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Endorse having low back pain as a primary or secondary pain problem in the past 6 months;
3. Meet criteria for having a chronic pain problem (≥3 months, with pain experienced on ≥50% of days in past 6 months);
4. Average intensity of chronic pain ≥3 on a 10-point scale for most days of the previous 3 months;
5. Chronic pain interference for general activities ≥3 on a 10-point scale for the past 3 months;
6. Able to read, speak, and understand English;
7. If currently taking analgesic or psychotropic medication, medications must have been stabilized for ≥4 weeks prior to this study; and
8. Availability of a telephone, webcam, and microphone through computer or telephone, as well as daily internet access.

Exclusion Criteria:

1. Primary pain condition is headache;
2. Severe cognitive impairment;
3. Current alcohol or substance dependence;
4. Active malignancy (e.g., cancer not in remission), terminal illnesses, or serious medical conditions that may interfere with either study participation or with receiving potential treatment benefits (e.g., severe lupus);
5. Inability to walk (defined as unable to walk at least 50 yards), which would limit the ability of participants to benefit from the activation skills intervention;
6. Significant pain from a recent surgery or injury;
7. Pain condition for which surgery has been recommended and is planned;
8. Any planned surgery, procedure, or hospitalization that may conflict with or otherwise influence participation in the study;
9. Currently receiving or had received other psychosocial treatments for any pain condition;
10. Current or past participation in a research study with treatment components that may overlap those in the current study;
11. Current or history of diagnosis of primary psychotic or major thought disorder within the past 5 years;
12. Psychiatric hospitalization within the past 6 months;
13. Psychiatric or behavioral conditions in which symptoms were unstable or severe within the past 6 months;
14. Any psychiatric or behavioral issues as noted in the medical record or disclosed/observed during self-report screening that would indicate participant may be inappropriate in a group setting; and
15. Presenting symptoms at the time of screening that would interfere with participation, specifically active suicidal or homicidal ideation with intent to harm oneself or others or active delusional or psychotic thinking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, Ph.D., Principal Investigator — University of Washington; Melissa Day, Ph.D., Principal Investigator — The University of Queensland
Locations (1):
- University of Washington, Ninth and Jefferson Building, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make available to interested researchers a data file containing de-identified data used for each published article at the time the article is accepted for publication. The data will be de-identified to remove any variables from which it would be possible to identify any individual participants. Specifically, we will create a data file that includes all variables used in the published article and a list of the variables in the data file (along with variable labels) and mail to investigators who request the data a copy of: (1) the published article (which will describe the source of the data); (2) the variable list/variable labels; and (3) a CD of the data set (as an SPSS.sav file). Note, though, even though any data files that we share will be stripped of identifiers prior to release for sharing, it remains possible those who access the data could potentially use deduction to identify participants with unusual characteristics or combinations of unusual characteristics.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data used for the analyses for any papers published will become available to interested researchers by request after that article is published. Those data will continue to be available for at least five years following the publication of the article.
Access Criteria: We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Day MA, Ehde DM, Burns J, Ward LC, Friedly JL, Thorn BE, Ciol MA, Mendoza E, Chan JF, Battalio S, Borckardt J, Jensen MP. A randomized trial to examine the mechanisms of cognitive, behavioral and mindfulness-based psychosocial treatments for chronic pain: Study protocol. Contemp Clin Trials. 2020 Jun;93:106000. doi: 10.1016/j.cct.2020.106000. Epub 2020 Apr 14. PMID 32302791
- [Result] Day MA, Ciol MA, Mendoza ME, Borckardt J, Ehde DM, Newman AK, Chan JF, Drever SA, Friedly JL, Burns J, Thorn BE, Jensen MP. The effects of telehealth-delivered mindfulness meditation, cognitive therapy, and behavioral activation for chronic low back pain: a randomized clinical trial. BMC Med. 2024 Apr 12;22(1):156. doi: 10.1186/s12916-024-03383-2. PMID 38609994
- [Derived] Day MA, Ward LC, Ehde DM, Mendoza ME, Phillips Reindel KM, Thorn BE, Bindicsova I, Jensen MP. Initial development and psychometric properties of the Therapist Quality Scale. Rehabil Psychol. 2024 Nov;69(4):326-334. doi: 10.1037/rep0000550. Epub 2024 Feb 15. PMID 38358711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified primarily via coding lists (i.e., sections of medical charts) of UW Medicine patients who had a low back pain diagnosis in their electronic medical record. Other recruitment strategies included the use of the UW Rehabilitation Medicine departmental research participant pool, posted flyers in pain and rehabilitation clinics, clinician referrals, news releases with the UW Newsroom, and a variety of national recruitment strategies.
Pre-assignment Details: Of the 1081 participants screened for eligibility, 100 could not be contacted, 78 declined participation, 494 did not meet screening criteria, and 12 were not recruited as the recruitment period had concluded. A total of 397 were then enrolled and commenced the baseline assessments. Of those, 302 completed at least 10/14 EMA surveys and also returned the activity monitor with overall wear compliance at 70% of time or higher, and these participants were then randomized to condition.
Period: Overall Study
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Started | 99 | 102 | 101
Completed | 86 | 88 | 89
Not Completed | 13 | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition | Total
Number analyzed (Participants) | 99 | 102 | 101 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (14.7) | 49.4 (14.7) | 51.0 (12.2) | 49.1 (14.0)
Sex/Gender, Customized [Number; unit: participants]
  Woman | 78 | 76 | 78 | 232
  Man | 18 | 21 | 18 | 57
  Transgender | 0 | 1 | 0 | 1
  Non-binary | 2 | 1 | 1 | 4
  Other/Unspecified | 1 | 3 | 4 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 83 | 72 | 75 | 230
  Black/African American | 4 | 8 | 8 | 20
  Latinx | 3 | 8 | 8 | 19
  Other/Unspecified | 9 | 14 | 10 | 33
Region of Enrollment [Number; unit: participants]
  United States | 99 | 102 | 101 | 302
PROMIS Pain Interference [Mean (Standard Deviation); unit: T-score] — The raw scores are converted to T-scores, which are standardized scores with a mean of 50 and a standard deviation of 10. Higher scores represent higher levels of pain interference.
  T-score | 66.6 (5.2) | 64.9 (5.4) | 66.4 (5.9) | 65.98 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Interference (Micro-level Change)
Description: Change in pain interference with different activities/aspects of life will be measured with five items from the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference item bank. Responses from each item will be summed for a total raw score from 5-25. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate more self-reported pain interference with different activities/aspects of life. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: Assessed via EMA twice daily during 4-week treatment period, early treatment (1-2 weeks) and late treatment (3-4 weeks) reported
Population: Intent to treat sample.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
scores on a scale
  Early treatment slope (assessed via EMA) | -1.34 (9.93) | -1.03 (5.68) | -0.50 (4.73)
  Late treatment slope (assessed via EMA) | -0.73 (6.67) | 0.01 (6.05) | -0.73 (6.29)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — We hypothesized negligible between condition differences, although within each condition, we hypothesized that each treatment would produce medium effect size improvements; p > .05, ANOVA

2. Primary Outcome: Change in Pain Interference (Macro-level Change)
Description: Change in pain interference with different activities/aspects of life will be measured with five items from the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference item bank. Responses from each item will be summed for a total raw score from 5-25. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate more self-reported pain interference with different activities/aspects of life. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat sample.
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Change from pre- to post-treatment (assessed over phone) | -5.0 (5.0) | -4.5 (6.4) | -5.6 (5.6)
  Change from pre- to 3 months post-treatment (assessed over phone) | -4.7 (5.5) | -3.4 (6.2) | -5.6 (6.2)
  Change from pre- to 6 months post-treatment (assessed over phone) | -4.1 (6.0) | -3.4 (6.2) | -5.6 (7.0)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

3. Secondary Outcome: Change in Pain Intensity (Micro-level)
Description: Change in pain intensity of chronic pain in general will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their pain intensity. Higher scores indicate higher levels of self-reported pain intensity. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
scores on a scale
  Early treatment slope (assessed via EMA) | -0.40 (2.00) | -0.26 (1.67) | -0.23 (1.18)
  Late treatment slope (assessed via EMA) | -0.17 (1.26) | 0.09 (1.74) | -0.04 (1.79)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

4. Secondary Outcome: Change in Mood (Micro-level)
Description: Change in mood will be assessed using the Positive and Negative Affect Schedule (PANAS). Total scores will range from 1-5 for each affect schedule. A higher positive affect sum score indicates more self-reported positive affect while a lower negative affect sum score indicates less self-reported negative affect. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
scores on a scale
  Positive Affect, early treatment slope (assessed via EMA) | 0.13 (1.01) | 0.06 (0.89) | 0.01 (0.71)
  Negative Affect, early treatment slope (assessed via EMA) | -0.19 (0.82) | -0.08 (0.96) | -0.13 (0.73)
  Positive Affect, late treatment slope (assessed via EMA) | 0.08 (0.67) | 0.08 (0.60) | 0.16 (0.62)
  Negative Affect, late treatment slope (assessed via EMA) | -0.14 (0.73) | 0.05 (0.70) | 0.11 (0.75)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

5. Secondary Outcome: Change in Physical Function
Description: Change in extent of physical function will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form-4A. Responses from each item will be summed to form a total raw score ranging from 4-20. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher levels (i.e., better) physical function. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Change from pre- to post-treatment (assessed over phone) | 1.6 (3.6) | 1.1 (3.4) | 2.1 (3.8)
  Change from pre- to 3 months post-treatment (assessed over phone) | 2.0 (4.3) | 1.2 (4.0) | 2.7 (4.2)
  Change from pre- to 6 months post-treatment (assessed over phone) | 1.9 (5.6) | 1.3 (5.2) | 2.5 (4.8)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

6. Secondary Outcome: Change in Sleep Quality
Description: Change in sleep quality will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form-4A. Responses from each item will be summed to form a total raw score ranging from 4-20. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate more self-reported sleep disturbance. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Change from pre- to post-treatment (assessed over phone) | -3.5 (7.1) | -1.7 (6.2) | -4.9 (6.8)
  Change from pre- to 3 months post-treatment (assessed over phone) | -3.5 (6.6) | -2.1 (7.1) | -4.3 (8.3)
  Change from pre- to 6 months post-treatment (assessed over phone) | -4.0 (7.3) | -3.4 (7.6) | -4.9 (9.4)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.01, ANOVA

7. Secondary Outcome: Change in Depression Severity
Description: Change in depression will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form-4A. Responses from each item will be summed to form a total raw score ranging from 4-20. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher self-reported levels of depression. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Change from pre- to post-treatment (assessed over phone) | -3.3 (7.0) | -2.6 (7.8) | -2.6 (6.7)
  Change from pre- to 3 months post-treatment (assessed over phone) | -2.4 (6.9) | -2.3 (8.2) | -2.0 (6.4)
  Change from pre- to 6 months post-treatment (assessed over phone) | -2.3 (7.7) | -2.2 (9.4) | -1.9 (7.4)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

8. Secondary Outcome: Change in Anxiety Severity
Description: Change in anxiety will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form-4A. Responses from each item will be summed to form a total raw score ranging from 4-20. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher self-reported levels of anxiety. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Change from pre- to post-treatment (assessed over phone) | -2.2 (7.1) | -2.1 (7.9) | -1.5 (7.2)
  Change from pre- to 3 months post-treatment (assessed over phone) | -1.4 (8.6) | -2.2 (9.0) | -0.4 (8.3)
  Change from pre- to 6 months post-treatment (assessed over phone) | -1.8 (8.4) | -1.4 (9.4) | 0.1 (8.9)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

9. Secondary Outcome: Change in Medication Use
Description: Change in opioid medication use will be assessed by asking participants to report use of opioid medications within the past 7 days. Participants will be asked to report medication name, quantity per dose (e.g., 50 mg), and number of medication doses taken in the past week. Researchers will calculate a morphine equivalent dose (MED) for opioid medications. Due to violation of assumptions of normality, the MED data was transformed into a categorical variable (no prescription, increase, decrease, no change).
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 85 | 87 | 89
Participants
  No prescription pre or post-treatment | 58 | 61 | 58
  No prescription pre or 3 months post-treatment: number analyzed (Participants) | 81 | 78 | 79
  No prescription pre or 3 months post-treatment | 53 | 53 | 49
  No prescription pre or 6 months post-treatment: number analyzed (Participants) | 78 | 72 | 80
  No prescription pre or 6 months post-treatment | 50 | 48 | 51
  Increase from pre- to post-treatment | 9 | 10 | 6
  Increase from pre- to 3 months post-treatment: number analyzed (Participants) | 81 | 78 | 79
  Increase from pre- to 3 months post-treatment | 13 | 12 | 9
  Increase from pre- to 6 months post-treatment: number analyzed (Participants) | 78 | 72 | 80
  Increase from pre- to 6 months post-treatment | 11 | 13 | 10
  Decrease from pre- to post-treatment | 6 | 13 | 12
  Decrease from pre- to 3 months post-treatment: number analyzed (Participants) | 81 | 78 | 79
  Decrease from pre- to 3 months post-treatment | 8 | 10 | 14
  Decrease from pre- to 6 months post-treatment: number analyzed (Participants) | 78 | 72 | 80
  Decrease from pre- to 6 months post-treatment | 10 | 10 | 10
  No change from pre- to post-treatment | 12 | 3 | 13
  No change from pre- to 3 months post-treatment: number analyzed (Participants) | 81 | 78 | 79
  No change from pre- to 3 months post-treatment | 7 | 3 | 7
  No change from pre- to 6 months post-treatment: number analyzed (Participants) | 78 | 72 | 80
  No change from pre- to 6 months post-treatment | 7 | 1 | 9
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — We hypothesized negligible between condition differences, although within each condition, we hypothesized that each treatment would produce a greater proportion of people decreasing their dose relative to those increasing their dose during treatment; p > .05, Chi-squared

10. Secondary Outcome: Change in Pain Intensity (Macro-level)
Description: Change in pain intensity of chronic pain in general will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their pain intensity. Higher scores indicate higher levels of self-reported pain intensity. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Change from pre- to post-treatment (assessed over phone) | -1.0 (1.8) | -1.2 (2.1) | -1.3 (1.9)
  Change from pre- to 3 months post-treatment (assessed over phone) | -0.9 (1.7) | -0.8 (1.9) | -1.4 (2.2)
  Change from pre- to 6 months post-treatment (assessed over phone) | -1.0 (1.9) | -1.0 (2.0) | -1.1 (2.0)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

11. Other Pre Specified Outcome: Change in Pain Catastrophizing (i.e., Cognitive Content Mechanism; Micro-level)
Description: Change in pain catastrophizing will be measured with items from the University of Washington (UW) Concerns About Pain (CAP) item bank. Responses from the CAP were summed for a total raw score. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher levels of catastrophizing. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
scores on a scale
  Early treatment slope (assessed via EMA) | -2.3 (7.96) | -1.30 (7.72) | -0.71 (5.96)
  Late treatment slope (assessed via EMA) | -1.55 (7.69) | -0.27 (7.34) | -0.07 (5.65)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

12. Other Pre Specified Outcome: Change in Non-Judgment (i.e., Cognitive Process Mechanism; Micro-level)
Description: Change in non-judgment will be measured with items from the Pain-Related Cognitive Process Questionnaire (PCPQ) Non-Judgmental Scale. When assessed via phone, the full 6-item scale will be used while only four items are used in the EMA. Items will be averaged for a mean score from 0-4. Higher mean PCPQ scores indicate higher frequencies of using the adaptive cognitive process of non-judgment in responding to pain. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
scores on a scale
  Early treatment slope (assessed via EMA) | 0.31 (0.77) | 0.18 (0.84) | 0.10 (0.72)
  Late treatment slope (assessed via EMA) | 0.10 (0.73) | 0.10 (0.79) | 0.05 (0.68)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

13. Other Pre Specified Outcome: Change in Activity Level (Actigraph, Vector Magnitude Average Counts)
Description: Change in activity level will be measured by an actigraphy device worn by the participant measuring activity level. In this study, we used the vector magnitude average counts variable, which is the average of all activity counts recorded per minute that the device was worn (i.e., it removes non-wear times from analysis). Higher activity counts indicate higher intensity activities that day; the minimum possible score (theoretically is zero, with no theoretical maximum score). Slopes were calculated by computing the linear regression slopes for the Actigraph collected activity counts.
Time Frame: Worn daily during 4-week treatment period, early treatment (baseline-2 weeks) and late treatment (2-4 weeks) reported
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: activity counts
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
activity counts
  Early Treatment (at baseline to 2 weeks) | -148064.01 (955190.23) | -2380.15 (569389.47) | -82046.98 (430455.44)
  Late Treatment (at 2 weeks to 4 weeks) | 26392.50 (962819.17) | -38711.02 (980492.69) | 64274.53 (573771.91)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

14. Secondary Outcome: Change in Mood (Macro-level)
Description: Change in mood will be assessed using the Positive and Negative Affect Schedule (PANAS). Responses from the positive affect items will be summed for a total positive score ranging from 5-25 while responses from the negative affect items will be separately summed for a total negative score ranging from 5-25. A higher positive affect sum score indicates more self-reported positive affect while a lower negative affect sum score indicates less self-reported negative affect. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Positive Affect, change from pre- to post-treatment (assessed over phone) | 1.5 (3.5) | 1.3 (3.0) | 1.6 (3.9)
  Negative Affect, change from pre- to post-treatment (assessed over phone) | -1.2 (3.2) | -0.8 (4.1) | -1.3 (3.3)
  Positive Affect, change from pre- to 3 months post-treatment (assessed over phone) | 1.4 (3.6) | 0.4 (3.4) | 1.0 (4.1)
  Negative Affect, change from pre- to 3 months post-treatment (assessed over phone) | -0.8 (3.4) | -0.5 (3.6) | -1.0 (3.0)
  Positive Affect, change from pre- to 6 months post-treatment (assessed over phone) | 0.7 (3.9) | 1.1 (3.2) | 0.8 (4.2)
  Negative Affect, change from pre- to 6 months post-treatment (assessed over phone) | -0.7 (3.8) | -0.5 (4.2) | -1.0 (3.9)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

15. Other Pre Specified Outcome: Change in Pain Catastrophizing (i.e., Cognitive Content Mechanism; Macro-level)
Description: Change in pain catastrophizing will be measured with items from the University of Washington (UW) Concerns About Pain (CAP) item bank. Responses from the CAP were summed for a total raw score. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher levels of catastrophizing. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Change from pre- to post-treatment (assessed over phone) | -7.12 (8.45) | -6.91 (9.85) | -8.28 (8.12)
  Change from pre- to 3 months post-treatment (assessed over phone) | -6.72 (9.32) | -4.70 (8.76) | -7.97 (9.48)
  Change from pre- to 6 months post-treatment (assessed over phone) | -5.47 (10.29) | -5.82 (9.59) | -6.56 (9.62)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

16. Other Pre Specified Outcome: Change in Non-Judgment (i.e., Cognitive Process Mechanism; Macro-level)
Description: Change in non-judgment will be measured with items from the Pain-Related Cognitive Process Questionnaire (PCPQ) Non-Judgmental Scale. When assessed via phone, the full 6-item scale will be used while only four items are used in the EMA. Items will be averaged for a mean score from 0-4. Higher mean PCPQ scores indicate higher frequencies of using the adaptive cognitive process of non-judgment in responding to pain. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: Collected via phone at pre-treatment, immediately post- the 4-week treatment period, and at 3- and 6-mos after Tx
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 99 | 102 | 101
change score on a scale
  Change from pre- to post-treatment (assessed over phone) | 0.43 (1.14) | 0.45 (1.19) | 0.48 (1.20)
  Change from pre- to 3 months post-treatment (assessed over phone) | 0.39 (1.01) | 0.35 (1.34) | 0.57 (1.04)
  Change from pre- to 6 months post-treatment (assessed over phone) | 0.36 (0.98) | 0.41 (1.24) | 0.46 (1.20)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p > .05, ANOVA

ADVERSE EVENTS:
Time Frame: All participants were monitored/assessed for adverse events from enrollment through study completion, which was an average of 9 months.
Description: Adverse events (AEs) were self-reported by participants and documented in an electronic regulatory event. The majority of AEs reported by participants were conveyed to researchers without prompt. AE monitoring occurred at the beginning of each treatment session with therapists asking if anyone had any negative effects attributed to the treatment. Any concerns that met the definition of an AE were documented. AEs were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/102 | 0/101
Serious Adverse Events (participants affected / at risk) | 5/99 | 9/102 | 11/101
Other Adverse Events (participants affected / at risk) | 48/99 | 43/102 | 52/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Therapy (CT) Condition (N=99) | Mindfulness Meditation (MM) Condition (N=102) | Behavioral Activation (BA) Condition (N=101)
Hospitalization for infection or illness (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) — Not study related
New cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Not study related
Hospitalization for surgery or procedure (Surgical and medical procedures) | 1 (1) | 2 (2) | 2 (2) — Not study related
Victim of assault (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Not study related
Hospitalization for mental health disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Not study related
Hospitalization for cardiac event (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) — Not study related
Hospitalization for adverse reaction to/complication during medical treatment (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) — Not study related
Hospitalization for symptoms of unknown cause (General disorders) | 0 (0) | 1 (1) | 0 (0) — Not study related
Hospitalization for pulmonary event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) — Not study related
Hospitalization for increased pain (General disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
Hospitalization for neurologic event (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) — Not study related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Therapy (CT) Condition (N=99) | Mindfulness Meditation (MM) Condition (N=102) | Behavioral Activation (BA) Condition (N=101)
Skin irritation from ActiGraph wear (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 5 (7)
Non-study related injury/accident (Injury, poisoning and procedural complications) | 8 (9) | 10 (11) | 7 (7) — Not study related
Worsening chronic pain symptoms (General disorders) | 6 (7) | 5 (5) | 8 (8) — Not study related
Symptoms of cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Not study related
Migraine or other neurological system symptoms (Nervous system disorders) | 6 (6) | 3 (3) | 6 (9) — Not study related
Underwent surgery or a medical procedure (Surgical and medical procedures) | 8 (8) | 10 (10) | 12 (12) — Not study related
Symptoms of multiple organ systems (General disorders) | 5 (5) | 3 (4) | 5 (5) — Not study related
Symptoms of a vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) — Not study related
New/worsening infection (Infections and infestations) | 5 (5) | 4 (4) | 4 (5) — Not study related
Symptoms of the GI region (Gastrointestinal disorders) | 5 (6) | 3 (3) | 5 (6) — Not study related
Respiratory symptoms/illness (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 8 (8) | 12 (14) — Not study related
New neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) — Not study related
Experienced allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — Not study related
Symptoms of a blood and lymphatic system disorder (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1) — Not study related
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) — Not study related
Delusional thinking (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Not study related
Psychological stress due to completing study assessments (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Victim of assault (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Not study related
Undisclosed reason to ER (General disorders) | 1 (1) | 0 (0) | 0 (0) — Not study related
Symptoms of the renal/urinary system (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (3) — Not study related
Symptoms of an immune system disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Not study related
Symptoms of an ear or labyrinth disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) — Not study related
Increased depressed mood, anxiety, or PTSD (Psychiatric disorders) | 0 (0) | 4 (5) | 5 (5) — Not study related
Discomfort from wearing ActiGraph (General disorders) | 2 (2) | 3 (3) | 2 (2)
Symptoms of an eye disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related

LIMITATIONS AND CAVEATS:
This RCT compared three active treatments and lacked an inert (e.g., treatment as usual) and/or attention (e.g., support group) control condition; therefore, the potential effects of time and non-specific factors cannot be accounted for.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03687762/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03687762/ICF_001.pdf